CLINICAL TRIAL: NCT06195241
Title: The Safety and Efficacy of DaxibotulinumtoxinA-Lanm for Benign Essential Blepharospasm and Hemifacial Spasm
Brief Title: Effects of DaxibotulinumtoxinA for Blepharospasm and Hemifacial Spasm
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-15151; 2023-IST-DAXI-000186 (Other: Revance Therapeutics)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Benign Essential Blepharospasm; Hemifacial Spasm
MeSH Terms: conditions — Benign essential blepharospasm; Hemifacial Spasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This will be a single-arm, crossover study, in which each patient is his/her own historical control using a 2:1 conversion ratio of Daxxify to Botox units.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Benign Essential Blepharospasm or Hemifacial Spasm (Experimental): Patients with either Benign Essential Blepharospasms or Hemifacial Spasms
  Interventions: Drug: DaxibotulinumtoxinA

INTERVENTIONS:
Drug: DaxibotulinumtoxinA — Patients with Benign Essential Blepharospasm (BEB) or Hemifacial spasms (HFS) will be treated with DaxibotulinumtoxinA-Lanm (Daxxify) using a 2:1 conversion rate of Daxxify to Botox.
  Other Names: Daxxify

SUMMARY:
The goal of this clinical trial is to test the effects of DaxibotulinumtoxinA-Lanm (Daxxify) in patients with benign essential blepharospasms (BEB) and hemifacial spasms (HFS). The main questions to answer:

1. Is there clinically significant difference (measured by Jankovic Rating Scale (JRS) score from base to peak efficacy) for patients with BEB and HFS treated with Daxxify?
2. What percentage of patients achieve a clinical response?

Participants historically treated with Botox for either BEB or HFS will be crossed over to Daxxify treatment in order to serve as their own control and examine the efficacy of Daxxify.

DETAILED DESCRIPTION:
This will be a single-arm, crossover study, in which each patient is their own historical control using a 2:1 conversion ratio of Daxxify to Botox units. Study participants will be selected through the electronic medical records of ophthalmologists at Montefiore Medical Center. Medical documentation on each patient will include information on age, sex, race, Benign Essential Blepharospasm (BEB) diagnosis year and duration, Hemifacial Spasms (HFS) diagnosis year and duration, and past treatments.

The immediate effects (desired or undesired) of Daxxify observed within 48-72 hours, will be defined as (1) complete relief of spasms (2) partial relief to a tolerable level (3) mild to moderate ocular irritation (4) ptosis.

Overall efficacy will be evaluated using the base to peak efficacy (recorded in changes to Jankovic Rating Scale (JRS) scores) and be defined as (1) excellent (resolution of signs and symptoms, only requiring injections > 5-6 months (2) moderate (improvement in signs and symptoms but requiring repeated injections within < 5 months (3) poor (no improvement in signs and symptoms).

Adverse side effects will be documented, and Daxxify will be discontinued in any patients who develop significant side effects that outweigh the benefits.

ELIGIBILITY:
Inclusion Criteria:

* Benign essential blepharospasm (BEB) or hemifacial spasm (HFS) as diagnosed by an ophthalmologist.
* No known neurologic or neuromuscular systematic medications.
* No history or surgical intervention for BEB or HFS.

Exclusion Criteria:

* Patients will be excluded if age < 18, are pregnant, non-willing, or with contra-indications to botulinum toxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Response based on the Jankovic Rating Scale | Prior to treatment at beginning of study
  Therapeutic response of Daxxify will be measured as the significant difference between the baseline to peak efficacy scores using the modified Jankovic rating scale (JRS). The JRS scale is a validated physician rating scale that consists of two subscales: blepharospasm (or hemifacial spasm) severity and blepharospasm (or hemifacial spasm) frequency. Each subscale is based on a 5-point scale ranging from 0-4, where 0 indicates no symptoms or frequency and 4 indicates the most severe or frequent symptoms. Overall scores will be reported as the sum of the two subscales of severity and frequency of symptoms and will range from 0-8. Basic descriptive statistics will be used to summarize and report therapeutic response. The Wilcoxon signed-ranked test will be used to analyze paired ordinal data gathered from the JRS scores.
Therapeutic Response based on the Jankovic Rating Scale | 1 month post-treatment
  Therapeutic response of Daxxify will be measured as the significant difference between the baseline to peak efficacy scores using the modified Jankovic rating scale (JRS). The JRS scale is a validated physician rating scale that consists of two subscales: blepharospasm (or hemifacial spasm) severity and blepharospasm (or hemifacial spasm) frequency. Each subscale is based on a 5-point scale ranging from 0-4, where 0 indicates no symptoms or frequency and 4 indicates the most severe or frequent symptoms. Overall scores will be reported as the sum of the two subscales of severity and frequency of symptoms and will range from 0-8. Basic descriptive statistics will be used to summarize and report therapeutic response. The Wilcoxon signed-ranked test will be used to analyze paired ordinal data gathered from the JRS scores.
Therapeutic Response based on the Jankovic Rating Scale | 3 months post-treatment
  Therapeutic response of Daxxify will be measured as the significant difference between the baseline to peak efficacy scores using the modified Jankovic rating scale (JRS). The JRS scale is a validated physician rating scale that consists of two subscales: blepharospasm (or hemifacial spasm) severity and blepharospasm (or hemifacial spasm) frequency. Each subscale is based on a 5-point scale ranging from 0-4, where 0 indicates no symptoms or frequency and 4 indicates the most severe or frequent symptoms. Overall scores will be reported as the sum of the two subscales of severity and frequency of symptoms and will range from 0-8. Basic descriptive statistics will be used to summarize and report therapeutic response. The Wilcoxon signed-ranked test will be used to analyze paired ordinal data gathered from the JRS scores.
Therapeutic Response based on the Jankovic Rating Scale | On a monthly basis after 3-month timepoint until symptom free, up to a maximum of 9 months
  Therapeutic response of Daxxify will be measured as the significant difference between the baseline to peak efficacy scores using the modified Jankovic rating scale (JRS). The JRS scale is a validated physician rating scale that consists of two subscales: blepharospasm (or hemifacial spasm) severity and blepharospasm (or hemifacial spasm) frequency. Each subscale is based on a 5-point scale ranging from 0-4, where 0 indicates no symptoms or frequency and 4 indicates the most severe or frequent symptoms. Overall scores will be reported as the sum of the two subscales of severity and frequency of symptoms and will range from 0-8. Basic descriptive statistics will be used to summarize and report therapeutic response. The Wilcoxon signed-ranked test will be used to analyze paired ordinal data gathered from the JRS scores.

SECONDARY OUTCOMES:
Waning of Effect | Prior to treatment at beginning of study
  Waning of effect will be assessed by quantifying the patient-reported time, in months, to noticing a loss of peak treatment effect. The number of months until noticing a loss of peak treatment effect will be summarized and reported using basic descriptive statistics.
Waning of Effect | 1 month post-treatment
  Waning of effect will be assessed by quantifying the patient-reported time, in months, to noticing a loss of peak treatment effect. The number of months until noticing a loss of peak treatment effect will be summarized and reported using basic descriptive statistics.
Waning of Effect | 3 months post-treatment
  Waning of effect will be assessed by quantifying the patient-reported time, in months, to noticing a loss of peak treatment effect. The number of months until noticing a loss of peak treatment effect will be summarized and reported using basic descriptive statistics.
Waning of Effect | On a monthly basis after 3-month timepoint until symptom free, up to a maximum of 9 months
  Waning of effect will be assessed by quantifying the patient-reported time, in months, to noticing a loss of peak treatment effect. The number of months until noticing a loss of peak treatment effect will be summarized and reported using basic descriptive statistics.
Loss of Efficacy | Prior to treatment at beginning of study
  Loss of efficacy will be assessed by quantifying the patient-reported time, in months, to noticing a complete loss of efficacy. The number of months to complete loss of efficacy will be summarized and reported using basic descriptive statistics.
Loss of Efficacy | 1 month post-treatment
  Loss of efficacy will be assessed by quantifying the patient-reported time, in months, to noticing a complete loss of efficacy. The number of months to complete loss of efficacy will be summarized and reported using basic descriptive statistics.
Loss of Efficacy | 3 months post-treatment
  Loss of efficacy will be assessed by quantifying the patient-reported time, in months, to noticing a complete loss of efficacy. The number of months to complete loss of efficacy will be summarized and reported using basic descriptive statistics.
Loss of Efficacy | On a monthly basis after 3-month timepoint until symptom free, up to a maximum of 9 months
  Loss of efficacy will be assessed by quantifying the patient-reported time, in months, to noticing a complete loss of efficacy. The number of months to complete loss of efficacy will be summarized and reported using basic descriptive statistics.
Incidence Rate of Treatment Failure | Up to four week post treatment
  Participant incidence rate of treatment failure will be measured as a lack of response or primary non-response (defined as a < 25% response from the first injection and subsequent injections of increasing dosages) to medication up to four weeks later for either benign essential blepharospasm or hemifacial spasm. Incidence rate of treatment failure will be defined as the percentage of participants who did not respond to treatment and will be summarized using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barmettler, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No